CLINICAL TRIAL: NCT06262555
Title: Novel Light Delivery Method for Performing Transbronchial Photodynamic Therapy Ablation to Treat Peripheral Lung Cancer: A Second Phase Pilot Study
Brief Title: Novel Light Delivery Method for Performing Transbronchial Photodynamic Therapy for Peripheral Lung Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taoyuan General Hospital (Other Government)
Responsible Party: Principal Investigator, Clinical Research Center, Chief of Thoracic Surgery Department, Taoyuan General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TYGH111061
Record Dates: First submitted 2024-01-30; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Lung Cancer; Lung Cancer Metastatic
Keywords: Photodynamic Therapy; Peripheral Lung Cancer; Trans-Bronchoscope Ablation
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Arm 1 (Experimental): Photophrin 2mg/kg 48 hours before treatment. Navigational bronchoscope guide the catheter into the tumor and adjacent to the tumor and give lipiodol for light diffusion and give light 200J/cm from different angle
  Interventions: Procedure: Transbronchial PDT peripheral lung tumor ablation

INTERVENTIONS:
Procedure: Transbronchial PDT peripheral lung tumor ablation — Transbronchial lung tumor ablation with Photodynamic therapy

SUMMARY:
This research aims to develop an innovative photodynamic therapy (PDT) for peripheral lung tumors. Current treatments involve surgery, chemotherapy, and radiation. Photodynamic therapy, using light and photosensitizing drugs, is promising but has limitations. Our team proposes using Lipiodol, a contrast agent, instilled into the trachea via bronchoscopy, surrounding the tumor. Preliminary pig model trials showed safety. Clinical trials, building on a U.S. study (NCT02916745), commenced in October 2021, treating three cases. Initial results suggest safety, but efficacy requires further investigation. Based on ongoing trials, we propose a phase I trial with multiple light treatments from different directions and an additional dose after 48 hours to assess safety and efficacy. This study will guide future clinical trials for optimal PDT dosage.

DETAILED DESCRIPTION:
The main focus of this research is the development of an innovative photodynamic therapy (PDT) mode applied to peripheral lung tumors. Current treatments for lung tumors, including primary lung cancer or metastatic tumors to the lungs, involve surgery, chemotherapy (including targeted and immunotherapy), and radiation therapy. The choice of treatment depends on factors such as tumor size, invasion, genetic characteristics, and the overall health of the patient.

For early-stage peripheral lung tumors, there is a continuous effort to develop minimally invasive treatment modalities to replace current surgical methods. Techniques such as computed tomography-guided percutaneous or bronchoscopic-guided radiofrequency ablation (RFA), microwave ablation, and photodynamic therapy are actively under research and development. Photodynamic therapy utilizes special photosensitizing drugs selectively absorbed by cancer cells, followed by exposure to light of specific wavelengths, triggering a reaction that destroys cancer cells.

Although photodynamic therapy has been successful in treating early-stage central airway lung cancer or advanced tumors causing airway obstruction, it has limitations. The penetration of light is restricted, resulting in a treatment range of approximately 1.5 to 2 centimeters in diameter. Multiple guidance and light treatments are needed to cover the entire tumor, increasing the technical difficulty of the procedure.

Light travels in a straight line and undergoes penetration, absorption, and reflection when encountering tissue interfaces, limiting its penetration within tissues. Dr. Friedberg in the United States proposed a novel lighting mode in 2003, using materials with high refractive indices, such as mineral oil (refractive index approximately 1.47), to enable light conduction in the trachea and bronchi. However, mineral oil is harmful to lung tissue, causing severe complications if inadvertently inhaled into the airways.

In this study, Lipiodol, a contrast agent with a refractive index of 1.47, was considered as a potential alternative to mineral oil. Lipiodol is a mixture of poppy seed oil and iodine ions and is commonly used in lymphography or for embolization therapy of liver tumors. It has been used for years in clinical practice for bronchoscopic instillation as a means of visualizing and locating lung tumors.

Based on these considerations, the research team hypothesized that by using electromagnetic navigation bronchoscopy to instill Lipiodol into the proximal trachea of the lung segment containing the tumor, the tumor could be completely surrounded by Lipiodol. Subsequent light therapy in the proximal trachea would then illuminate the lung tissue containing Lipiodol, including the tumor tissue, supplying blood vessels, and lymphatic tissue, selectively killing tumor tissue and potential early micro-metastases.

The research team conducted preclinical trials using a pig model, confirming that Lipiodol could be instilled into the peripheral lung tumor location via bronchoscopy. Moreover, light therapy with the current energy settings (200 J/cm, 400 mW/cm, 500 seconds) in Lipiodol-injected lung tissue was shown to be safe.

A multi-center clinical trial in the United States (ClinicalTrials.gov Identifier: NCT02916745) explored PDT for peripheral lung tumors. Photofrin was intravenously injected 48 hours before treatment, and under the guidance of electromagnetic navigation bronchoscopy and bronchoscopic ultrasound, the light fiber was inserted into the tumor site for PDT with an energy setting of 200 J/cm, 400 mW/cm, 500 seconds. The trial, as of January 2019, included five patients with no reports of severe complications, indicating initial safety and feasibility. Building upon this trial and the team's proposed novel PDT lighting mode, a phase I human clinical trial was initiated in October 2021 and is ongoing until February 2022. Three cases have been treated, and the initial observations suggest safety and feasibility. One patient, unfortunately, succumbed to obstructive pneumonia six weeks after treatment due to rapid disease progression, but it was not considered a treatment-related complication.

Although the effectiveness of the treatment was not as anticipated, further clinical trials are needed to determine the optimal lighting dosage. In the ongoing trial (NCT02916745), two cases received multiple light treatments from different directions without significant complications. A case report by Dr. Allison demonstrated successful and complication-free bronchoscopic PDT with two light treatments 48 hours apart in a patient ineligible for standard treatments.

The next phase of clinical trials is proposed based on the team's 2022 single-light treatment trial, aiming to assess safety and efficacy using multiple light treatments in different directions and an additional dose 48 hours later. This study will serve as a reference for the minimum basic lighting dosage (NOAEL) and the possible effective dosage for future phase I clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with advanced or terminal malignant lung tumors (including primary lung cancer and lung metastases from other cancers).
* Patients who have failed standard treatments (surgery, radiotherapy, or first and second-line chemotherapy/immunotherapy/targeted therapy) or are unsuitable for standard treatments.
* Tumor size less than or equal to 3 cm, clearly assessable on chest computed tomography.

Patients capable of providing informed consent and willing to undergo regular follow-ups during the trial.

Exclusion Criteria:

* Diagnosis of small cell lung cancer or non-solid malignancies.
* Tumors located in the central part of the lungs.
* Previous radiation therapy to the treatment site.
* Abnormal blood biochemical values.
* Chemotherapy received within the past 4 weeks.
* Tumor invading major blood vessels.
* Allergy to porphyrins or porphyrin-related metabolites, or allergy to Lipiodol or iodine-containing contrast agents.
* Planning radical surgery for lung tumors within the next 90 days.
* Potential need for slit lamp ophthalmic examination within the next 30 days due to existing eye diseases.
* Inability to undergo bronchoscopy due to mental health conditions.
* Pregnancy, planning pregnancy, breastfeeding, or planning to breastfeed within the next 6 months.
* Previous photodynamic therapy within the past 1 month.
* Severe kidney or liver disease with abnormal function.
* Planning to participate in other cancer treatment clinical trials within the next 3 months.
* HIV-positive patients.
* Individuals deemed unsuitable for the trial by the principal investigator and the safety monitoring committee due to severe illnesses.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Technical Feasibility | 3 days
  Number of times photodynamic therapy was delivered into the tumor using navigational bronchoscopy for each subject
Technical Safety | 6 months
  Events Incidence Indicating Safety of Novel Photodynamic Therapy The incidence of adverse events following Novel PDT will be presented as the primary safety indicator for this treatment.

SECONDARY OUTCOMES:
Tumor remission rate | 3 months
  Tumor Response at 3 Months Post Photodynamic Therapy (PDT) From the start of treatment until 6 months post-treatment measured as per the Modified RECIST (Response Evaluation Criteria in Solid Tumors) Criteria

CONTACTS AND LOCATIONS:
Overall Officials: Yei San Hsieh, Principal Investigator — Taoyuan General Hospital
Locations (1):
- Taoyuan General Hospital, Ministry of Health and Welfare, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided